CLINICAL TRIAL: NCT01669044
Title: Comparison the Hemodynamics Effects Between Dexmedetomidine and Propofol in Major Abdominal Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Minying Chen, MD, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: IRB[2012]260
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Abdominal Tumor; Intestinal Obstruction; Cirrhosis; Intestinal Fistula; Aneurism
MeSH Terms: conditions — Abdominal Neoplasms; Intestinal Obstruction; Fibrosis; Intestinal Fistula | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- dexmedetomidine,hemodynamics,injection: Group 1:when the patient can be roused after major abdominal surgery ，we will inject dexmedetomidine at 1μg/kg in 10 minutes as a loading dose, followed by a continuous infusion at 0.3μg/kg/h for 6 to 24hours.then adjust the infusion dose to maintain the ramsay scale at 3-4 scores.
  Interventions: Drug: dexmedetomidine
- propofol,hemodynamics,injection: Group 2 :when the patient can be roused after major abdominal surgery ，we will inject propofol at 0.5mg/kg as a loading dose, followed by a continuous infusion at 0.5mg/kg.h for 6 to 24hours.then adjust the infusion dose to maintain the ramsay scale at 3-4 scores
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: dexmedetomidine — dexmedetomidine: IV (in the vein)at 1μg/kg in 10 minutes as a loading dose, followed by a continuous infusion at 0.3μg/kg/h.then adjust the infusion dose to maintain the ramsay scale at 3-4 scores.
  Groups: dexmedetomidine,hemodynamics,injection
Drug: propofol — propofol: IV (in the vein)at 0.5mg/kg as a loading dose, followed by a continuous infusion at 0.5mg/kg/h.then adjust the infusion dose to maintain the ramsay scale at 3-4 scores.
  Groups: propofol,hemodynamics,injection

SUMMARY:
The alpha2 agonist dexmedetomidine is a new sedative agent combined with the analgesic qualities and lack of respiratory depression. Patients sedated with dexmedetomidine could be easily roused, these advances shows dexmedetomidine may be a effective and safe sedative agent. But some studies showed some adversely effects of dexmedetomidine on haemodynamics (such as bradycardia, hypotension), the investigators want to further research the effects of dexmedetomidine on haemodynamics, such as Cardiac Output (CO), Systemic Venous Resistance Index(SVRI), and so on. Propofol is widely used sedative agent in ICU, it also has adversely effects like bradycardia and hypotension, so the investigators want to compare the effect of dexmedetomidine with propofol on haemodynamics after major abdominal surgery. Expect to further research the mechanism of haemodynamics of dexmedetomidine.

DETAILED DESCRIPTION:
When the patients can be roused, they will first receive analgesia with bolus of fentanyl 0.03mg, followed by a continuous infusion at a ﬁxed dose of 0.3μg/kg/h during study period. Then patients will be randomly divided into two groups (Dexmedetomidine and Propofol). All of them will receive hemodynamic monitoring through "Vigileo"(Edwards Lifesciences) and cardiogram monitor. The study will continue for 6-24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Postoperative patients of major abdominal surgery
2. Age ≧ 18

Exclusion Criteria:

1. heart rate ≤ 50 bpm
2. allergy with dexmedetomidine or propofol
3. pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postoperative patients of major abdominal surgery
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2012-05; Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Cardiac output | the study will start when the patient can be roused after major abdominal surgery and will continue for 6 to 24hours

SECONDARY OUTCOMES:
Stroke Volume | the study will start when the patient can be roused after major abdominal surgery and will continue for 6 to 24hours

OTHER OUTCOMES:
Systemic Venous Resistance Index | the study will start when the patient can be roused after major abdominal surgery and will continue for 6 to 24hours

CONTACTS AND LOCATIONS:
Overall Officials: minying chen, MD, Principal Investigator — study principal investigator
Locations (1):
- First affiliated hostipal,Sun Yat-sen University, Guangzhou, Guangdong, China